CLINICAL TRIAL: NCT02072096
Title: An Individualized treatMent aPproach for oldER patIents: A Randomized, Controlled stUdy in Type 2 Diabetes Mellitus (IMPERIUM)
Brief Title: A Comparison of Two Treatment Strategies in Older Participants With Type 2 Diabetes Mellitus (T2DM)
Acronym: IMPERIUM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was terminated per protocol because of lack of feasibility.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14842; F3Z-MC-IOQL (Other: Eli Lilly and Company); 2013-001473-24 (EudraCT Number)
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Metformin; Pioglitazone; Acarbose; Linagliptin; Sitagliptin Phosphate; Liraglutide; Insulin Glargine; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strategy A (Glucose-Dependent) (Experimental): Participants may receive oral and injectable (glucagon-like peptide-1 receptor agonists [GLP-1 RA]) therapies that exert a glucose-dependent mode of action. Medications allowed in this arm include: metformin, pioglitazone, acarbose, linagliptin, sitagliptin, liraglutide, exenatide once weekly (QW), and exenatide twice daily (BID). Choice of therapy is based on investigator's discretion. Treatment used in label. Treatment may last up to 72 weeks.
  Interventions: Drug: Metformin; Drug: Pioglitazone; Drug: Acarbose; Drug: Linagliptin; Drug: Sitagliptin; Drug: Liraglutide; Drug: Exenatide once weekly (QW); Drug: Exenatide twice daily (BID)
- Strategy B (Reference) (Active Comparator): Participants will receive glimepiride and may receive basal insulin glargine as a first line injectable therapy. Medications allowed in this arm include: glimepiride, metformin, pioglitazone, acarbose, linagliptin, sitagliptin and basal insulin glargine. Choice of therapy is based on investigator's discretion. Treatment used in label. Insulin glargine is titrated according treatment algorithm. Treatment may last up to 72 weeks.
  Interventions: Drug: Glimepiride; Drug: Metformin; Drug: Pioglitazone; Drug: Acarbose; Drug: Linagliptin; Drug: Sitagliptin; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Glimepiride — Administered orally
  Arms: Strategy B (Reference)
Drug: Metformin — Administered orally
Drug: Pioglitazone — Administered orally
Drug: Acarbose — Administered orally
Drug: Linagliptin — Administered orally
Drug: Sitagliptin — Administered orally
Drug: Liraglutide — Administered subcutaneously (SC)
  Arms: Strategy A (Glucose-Dependent)
Drug: Insulin Glargine — Administered SC
  Arms: Strategy B (Reference)
Drug: Exenatide once weekly (QW) — Administered SC
  Arms: Strategy A (Glucose-Dependent)
Drug: Exenatide twice daily (BID) — Administered SC
  Arms: Strategy A (Glucose-Dependent)

SUMMARY:
The main purpose of this study is to compare the benefits and risks associated with the use of 2 treatment strategies to lower blood sugar in participants aged 65 and older with T2DM. One strategy is based on the use of oral and injectable medications that only reduce blood sugar (glucose) when it is high. The other strategy is based on non-glucose dependent agents. The trial will last up to 72 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have T2DM based on a history and clinical impression that is consistent with the World Health Organization (WHO) Classification of Diabetes
* Have a Clinical Frailty Scale (CFS) score of 4 or above or Total Illness Burden Index (TIBI) score of 5 or above as assessed at screening
* Have an A1c >7.3% and <10.9% at study entry and are not achieving desired glycemic control as evidenced by A1c measurement at least 0.4% higher than individualized treatment target set at screening.
* Have been treated for at least 3 months prior to the study entry with any of the following treatment options:

  * Diet/exercise only (only if they have known contraindications to metformin treatment)
  * Any dose of sulfonylurea
  * Effective or maximally-tolerated doses of metformin, dipeptidyl-peptidase-4 (DPP-4) inhibitor, thiazolidinedione, or acarbose used in monotherapy or in dual combination. The following doses are considered to be effective:

    * at least 1500 mg of metformin per day
    * At least 30 mg of pioglitazone per day
    * At least 4 mg of rosiglitazone per day
    * At least 75 mg of acarbose per day
    * Any marketed dose of DPP-4 inhibitor

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving an investigational product or nonapproved use of a drug or device (other than the investigational product used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated, within the last 60 days in a clinical trial involving an investigational product other than the investigational product used in this study. If the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed
* Have previously completed or withdrawn from this study. This exclusion criterion does not apply to participants who are rescreened prior to randomization
* At study entry, have contraindications to sulfonylurea, insulin, or GLP-1 RA
* Have a history of pancreatitis, a personal or family history of medullary thyroid carcinoma, or have Multiple Endocrine Neoplasia syndrome type 2
* Have taken any injectable glucose-lowering agent, miglitol, meglitinide, Sodium/Glucose cotransporter-2 inhibitor, or other antihyperglycemia treatment that is not listed in the fourth inclusion criterion for more than 10 days within 3 months prior to the study entry
* In the opinion of investigator should have an individualized A1c target set at 8% or higher
* Have a body mass index (BMI) greater than 45 kg/m^2
* Have had more than 1 episode of severe hypoglycemia within 24 weeks prior to the study
* Have cardiac disease with functional status that is Class III or IV according to the New York Heart Association Cardiac Disease Classification
* Have an estimated glomerular filtration rate (eGFR) <30 milliliter/minute/1.73 m^2 (mL/min/1.73 m^2) or advanced renal disease including history of renal transplantation or currently receiving renal dialysis
* Have obvious clinical signs or symptoms or laboratory evidence of liver disease (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] > 2.5 times the upper limit of the reference range)
* Receive current therapy for a malignancy, other than basal-cell or squamous-cell skin cancer
* Received systemic glucocorticoids within the 3 months prior to entry for more than 14 consecutive days
* Have any other condition that precludes the participant from following and completing the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 192 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (33):
- United States (16):
  - Suncoast Research Group, LLC, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Florida Hospital, Orlando, Florida
  - Athens Primary Care, Athens, Georgia
  - Herman Clinical Research, LLC, Suwanee, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Iderc, P.L.C., Des Moines, Iowa
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Mercy Health Research, St Louis, Missouri
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Family Medical Associates, Levittown, Pennsylvania
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Rockwood Clinic Research Center, Spokane, Washington
- Austria (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Stefan Ob Stainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salzburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dortmund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuwied
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stuttgart
- Puerto Rico (2):
  - Manati Medical Center, Manatí
  - American Telemedicine Center, San Juan
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salford, Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dundee, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sheffield, South Yorkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ipswich, Suffolk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Heller SR, Pratley RE, Sinclair A, Festa A, Kiljanski J, Brusko CS, Duan R, Heine RJ. Glycaemic outcomes of an Individualized treatMent aPproach for oldER vulnerable patIents: A randomized, controlled stUdy in type 2 diabetes Mellitus (IMPERIUM). Diabetes Obes Metab. 2018 Jan;20(1):148-156. doi: 10.1111/dom.13051. Epub 2017 Aug 8. PMID 28671753

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed the first 24 weeks of the study at which time the study was stopped and interim analysis was triggered to assess feasibility. Treatment continued per protocol until study termination and participants discontinued at the next office study visit. Data was assessed from Baseline to last participant visit, up to 72 weeks.
Groups:
- Strategy A (Glucose-Dependent): Participants may receive oral and injectable therapies (glucagon-like peptide-1 receptor agonists [GLP-1 RA]) that exert a glucose-dependent mode of action. Medications allowed in this arm include: metformin, pioglitazone, acarbose, linagliptin, sitagliptin, liraglutide, exenatide once weekly (QW), and exenatide twice daily (BID). Choice of therapy is based on investigator's discretion. Treatment used in label. Treatment may last up to 72 weeks.
- Strategy B (Reference): Participants will receive glimepiride and may receive basal insulin glargine as a first line injectable therapy. Medications allowed in this arm include: glimepiride, metformin, pioglitazone, acarbose, linagliptin, sitagliptin and basal insulin glargine. Choice of therapy is based on investigator's discretion. Treatment used in label. Insulin glargine is titrated according to treatment algorithm. Treatment may last up to 72 weeks.
Period: Overall Study
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference)
Started | 99 | 93
Received at Least One Dose of Study Drug | 98 | 93
Completed | 14 | 15
Not Completed | 85 | 78
Not completed — Lack of Efficacy | 18 | 29
Not completed — Protocol Violation | 7 | 7
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Adverse Event | 5 | 2
Not completed — No Reason Provided | 4 | 2
Not completed — Death | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Study Terminated by Sponsor | 43 | 30
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Strategy B (Reference): Participants will receive glimepiride and may receive basal insulin glargine as a first line injectable therapy. Medications allowed in this arm include: glimepiride, metformin, pioglitazone, acarbose, linagliptin, sitagliptin and basal insulin glargine. Choice of therapy is based on investigator's discretion. Treatment used in label. Insulin glargine dose is titrated according to treatment algorithm. Treatment may last up to 72 weeks.
- Total: Total of all reporting groups
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference) | Total
Number analyzed (Participants) | 99 | 93 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (5.3) | 70.7 (4.4) | 70.7 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 34 | 77
  Male | 56 | 59 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 32 | 67
  Not Hispanic or Latino | 63 | 59 | 122
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 93 | 81 | 174
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 18 | 14 | 32
  Puerto Rico | 23 | 16 | 39
  United States | 29 | 35 | 64
  United Kingdom | 10 | 11 | 21
  Germany | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving and Maintaining Individualized Glycated Hemoglobin A1c (HbA1c) Targets Without Clinically Significant Hypoglycemia
Description: Failed to reach and maintain HbA1c target, without clinically significant hypoglycemia, is defined as having 2 consecutive HbA1c > upper limit of HbA1c target over 12 weeks starting from Week 24 for participants with HbA1c data beyond Week 24, or Week 24 HbA1c > upper limit of HbA1c target for participants without HbA1c data beyond Week 24. Clinically significant hypoglycemia is defined as any severe hypoglycemia or repeated hypoglycemia interrupting participants activities or sleep and associated with blood glucose ≤3.9 millimole per liter (mmol/L), or repeated asymptomatic hypoglycemia associated with blood glucose <3.0 mmol/L. Success is defined as lacking of failure.
Time Frame: Baseline to last participant visit (up to 72 weeks)
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Strategy B (Reference): Participants will receive glimepiride and may receive basal insulin glargine as a first line injectable therapy. Medications allowed in this arm include: glimepiride, metformin, pioglitazone, acarbose, linagliptin, sitagliptin and basal insulin glargine. Choice of therapy is based on investigator's discretion. Treatment used in label. Dose titrated by treatment algorithm. Treatment may last up to 72 weeks.
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference)
Number analyzed (Participants) | 98 | 93
percentage of participants | 64.5 [54.4 to 73.4] | 54.9 [44.6 to 64.9]

2. Secondary Outcome: Percentage of Participants Requiring Alternative Treatment Due to Glycemic Failure of First Line Injectable Therapy
Time Frame: Baseline to last participant visit (up to 72 weeks)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference)
Number analyzed (Participants) | 98 | 93
percentage of participants | 21 | 13

3. Secondary Outcome: Number of Participants With Total Hypoglycemia and Other Categories of Hypoglycemia
Time Frame: Baseline to last participant visit (up to 72 weeks)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference)
Number analyzed (Participants) | 98 | 93
Participants
  Total Hypoglycemia | 10 | 50
  Severe Hypoglycemia | 0 | 0
  Clinically Significant Hypoglycemia | 0 | 1
  Symptomatic Hypoglycemia | 5 | 34
  Asymptomatic Hypoglycemia | 8 | 30
  Probable Symptomatic Hypoglycemia | 0 | 7
  Unspecified Hypoglycemia | 2 | 7
  Relative Hypoglycemia | 1 | 6
  Nocturnal Hypoglycemia | 4 | 10

4. Secondary Outcome: Change From Baseline of Urinary Albumin to Creatinine Ratio
Description: The Urinary Albumin to Creatinine Ratio is used in addition to Estimated Glomerular Filtration Rate (eGFR) to measure the incidence and progression of diabetic kidney disease.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had evaluable baseline and post-baseline urinary albumin to creatinine ratio.
Measure: Mean (Standard Deviation); unit: milligram per millimole (mg/mmol)
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference)
Number analyzed (Participants) | 80 | 83
milligram per millimole (mg/mmol) | 1.85 (22.99) | 1.85 (16.46)

5. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had evaluable baseline and post-baseline BMI data.
Measure: Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)
Groups:
- Strategy A (Glucose-Dependent): Participants may receive oral and injectable therapies (glucagon-like peptide-1 receptor agonists [GLP-1 RA]) that exert a glucose-dependent mode of action. Medications allowed in this arm include: metformin, pioglitazone, acarbose, linagliptin, sitagliptin, liraglutide, exenatide once weekly (QW), and exenatide twice daily (BID). Choice of therapy is based on investigator's discretion. Treatment used in label.Treatment may last up to 72 weeks.
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference)
Number analyzed (Participants) | 96 | 93
kilogram per square meter (kg/m^2) | -0.47 (1.56) | 0.20 (2.91)

6. Secondary Outcome: Change From Baseline of Estimated Glomerular Filtration Rate (eGFR)
Description: The eGFR is used in addition to the Urinary Albumin to Creatinine Ratio to measure the incidence and progression of diabetic kidney disease.
Time Frame: Baseline, Week 72
Population: All participants who received at least one dose of study drug and had evaluable baseline and post-baseline eGFR data.
Measure: Mean (Standard Deviation); unit: milliliter per minute/1.73 square meter
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference)
Number analyzed (Participants) | 85 | 85
milliliter per minute/1.73 square meter | -5.00 (13.64) | -5.88 (10.95)

7. Other Pre Specified Outcome: Change From Baseline in Adult Low Blood Sugar Survey (ALBSS) Score
Time Frame: Baseline, Week 72
Population: Unable to conduct change from baseline analysis due to study closure and lack of endpoint data.
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference)
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Change From Baseline in European Quality of Life-5 Dimensions 5 Levels (EQ-5D-5L) Score
Time Frame: Baseline, Week 72
Population: Unable to conduct change from baseline analysis due to study closure and lack of endpoint data.
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference)
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Change From Baseline in Mini-mental State Examination (MMSE) Score
Time Frame: Baseline, Week 72
Population: Unable to conduct change from baseline analysis due to study closure and lack of endpoint data.
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug.
Arm/Group | Strategy A (Glucose-Dependent) | Strategy B (Reference)
Serious Adverse Events (participants affected / at risk) | 15/98 | 14/93
Other Adverse Events (participants affected / at risk) | 82/98 | 74/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strategy A (Glucose-Dependent) (N=98) | Strategy B (Reference) (N=93)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Retinal vascular thrombosis (Eye disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strategy A (Glucose-Dependent) (N=98) | Strategy B (Reference) (N=93)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Type v hyperlipidaemia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 2 (2) | 3 (3)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Primary hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 12 (18) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (4) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 3 (3)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (5) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (3) | 2 (2)
Injection site nodule (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 6 (7) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 6 (6)
Peripheral swelling (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (2)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 4 (6) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chikungunya virus infection (Infections and infestations) | 4 (4) | 5 (5)
Colon gangrene (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 2 (2) | 0 (0)
Gingivitis (Infections and infestations) | 2 (3) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 3 (3)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (17) | 16 (18)
Onychomycosis (Infections and infestations) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 2 (2)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 7 (7)
Urinary tract infection (Infections and infestations) | 3 (3) | 8 (9)
Viral infection (Infections and infestations) | 2 (2) | 2 (2)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 4 (5)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (2) | 4 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriogram coronary (Investigations) | 0 (0) | 1 (2)
Arthroscopy (Investigations) | 2 (2) | 0 (0)
Aspiration pleural cavity (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose abnormal (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 2 (2) | 1 (1)
Blood pressure diastolic decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 1 (1)
Blood pressure systolic decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 1 (1) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Blood uric acid (Investigations) | 1 (1) | 0 (0)
Cardiac imaging procedure (Investigations) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 5 (5) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fructose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 9 (9) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 11 (11)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 7 (14) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Food aversion (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (2) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (5)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 3 (3) | 2 (4)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Lens extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Ptosis repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Tendon sheath lesion excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 1 (3)
Hypertension (Vascular disorders) | 5 (5) | 4 (5)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 2 (2)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated per protocol due to lack of feasibility. All participants completed the first 24 weeks of the study. Some participants continued into the Core study. Data was assessed from Baseline to last participant visit, up to 72 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No